CLINICAL TRIAL: NCT05650138
Title: Effects of Jacobson's Progressive Muscular Relaxation Technique on Blood Pressure Regulation and Activity of Daily Living in Hypertensive Patients
Brief Title: Effects of Jacobson's Progressive Muscular Relaxation Technique in Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0338
Record Dates: First submitted 2022-11-08; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Hypertension
Keywords: Hypertension; blood pressure; Relaxation; PMR
MeSH Terms: conditions — Hypertension | interventions — Walking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- jacobson's progressive muscular relaxation technique (Experimental): Questionnaire will be used as subjective measurements of activity of daily living and Bp will be monitored for initial readings. They will receive Jacobsons muscle relaxation technique. Patients will be demonstrated with the technique to contract and relax various groups of muscles, to coordinate contractions and relaxations with deep breaths and to perform the entire procedure with eyes closed in supine lying down position. Every subject will perform this supervised relaxation for 6 repetitions during a single session on once a day basis twice a week for four weeks. At the end of 4 weeks of treatment session blood pressure will be recorded questionnaire will be filled
  Interventions: Other: Jacobson's progressive muscular relaxation technique; Other: 30 min walk
- 30 min walk (Active Comparator): 4 weeks, twice a week, 30 minutes walk
  Interventions: Other: 30 min walk

INTERVENTIONS:
Other: Jacobson's progressive muscular relaxation technique — subjects will receive Jacobsons muscle relaxation technique. Patients will be demonstrated with the technique to contract and relax various groups of muscles, to coordinate contractions and relaxations with deep breaths and to perform the entire procedure with eyes closed in supine lying down position. Every subject will perform this supervised relaxation for 6 repetitions during a single session on once a day basis for four weeks.
  Arms: jacobson's progressive muscular relaxation technique
Other: 30 min walk — 30 minutes walk twice a week for 4 weeks

SUMMARY:
Effects of Jacobson's progressive muscular relaxation technique on blood pressure regulation and activity of daily living in hypertensive patient

DETAILED DESCRIPTION:
Hypertension is a disease that becomes a major problem of health. In 2008, 40% of adults aged 25 years above were diagnosed with hypertension. The mortality rate of the complications of hypertension reaches 9.4 million deaths worldwide each year. Hypertension is often called a ''silent killer'' because it often appears without symptoms until it becomes severe and impacts on other organs. Hypertension affects both on physical and psychological. Several studies have found that hypertension can cause anxiety. Hypertension requires comprehensive pharmacological and non-pharmacological treatment. Since 1983, the World Health Organization has suggested the use of the non-pharmacological approach in hypertension treatment. Progressive Muscle Relaxation (PMR) is one of the therapies that is mostly used in complementary therapy and alternative medication. PMR is a technique developed by Edmund Jacobson in 1920. This technique is designed to create a state of physiological and psychological relaxation in patients. It requires the patient to tense and relax various muscle groups while focusing awareness on proprioceptive and interceptive sensations. Several studies have found that PMR exercise helps to reduce blood pressure. Besides, PMR exercise can also reduce anxiety in various diseases.

Study design will be randomized controlled trial. Study will be conducted at Life care Hospital Gujranwala. Written informed consent will be obtained. Patients will be allocated randomly. Subjects meeting the predetermined inclusion and exclusion criteria . Questionnaire will be used as subjective measurements of activity of daily living and Bp will be monitored for initial readings.subjects will be divided into two groups both groups will perform 30 minutes walk as baseline treatment. only one group will receive Jacobsons muscle relaxation technique. Patients will be demonstrated with the technique to contract and relax various groups of muscles, to coordinate contractions and relaxations with deep breaths and to perform the entire procedure with eyes closed in supine lying down position. Every subject will perform this supervised relaxation for 6 repetitions during a single session on once a day basis for four weeks. At the end of 4 weeks of treatment session blood pressure will be recorded questionnaire will be filled. The data thus obtained will be considered for statistical analysis

ELIGIBILITY:
Inclusion Criteria:

* Age: 35 to 55 years
* Ambulatory male and female
* Mentally fitted
* Diagnosed with grade 2 and grade 3 hypertension(3)

Exclusion Criteria:

* Subjects who are not regular in taking medications and who reported about aggravation of any symptoms due to exercise.(7)
* Subjects who fall in grade1 hypertension
* Subjects below the age of 30.
* History of cardiac, renal and liver diseases
* History of recent fracture or surgery.

Ages: 33 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
changes in blood pressure | twice a week for four weeks
  subjects will receive Jacobsons muscle relaxation technique. Patients will be demonstrated with the technique to contract and relax various groups of muscles, to coordinate contractions and relaxations with deep breaths and to perform the entire procedure with eyes closed in supine lying down position. Every subject will perform this supervised relaxation for 6 repetitions during a single session on once a day basis for four weeks.
Barthel Index for Activity of daily living | four weeks
  The Barthel Index (BI) measures the extent to which somebody can function independently and has mobility in their activities of daily living feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing.

CONTACTS AND LOCATIONS:
Overall Officials: Sumera Abdulhameed, MS, Principal Investigator — Riphah International University
Locations (1):
- Life Care Hospital, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No